CLINICAL TRIAL: NCT02730949
Title: A Pilot Study of D-Chiro-Inositol Plus Folic Acid in Overweight Patients With Type 1 Diabetes
Brief Title: D-chiro-Inositol in Overweight Type 1 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Professor Paolo Pozzilli, Prof, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/14PARComETCBM
Record Dates: First submitted 2016-03-25; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
Keywords: D-Chiro-Inositol, type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 g D-chiro-Inositol + 400 mcg Folic Acid (Experimental): 1 g D-chiro-Inositol + 400 mcg folic acid once daily
  Interventions: Dietary Supplement: D-chiro-inositol; Dietary Supplement: Folic Acid
- 400 mcg folic (Active Comparator): 400 mcg folic acid only once daily
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: D-chiro-inositol — Treated group
  Arms: 1 g D-chiro-Inositol + 400 mcg Folic Acid
Dietary Supplement: Folic Acid — Control group

SUMMARY:
The purpose of this pilot study was to evaluate the effect of D-chiro-Inositol (DCI) oral supplementation in addiction to folic acid compared to folic acid alone on glycaemic control as assessed by HbA1c in overweight or obese T1D patients undergoing intensive insulin therapy.

A 24 weeks, prospective, randomized control trial was carried out in T1D patients, aged 17-50 years (13 males, 13 females), with disease duration > 1 year and BMI >25, attending as outpatients the Endocrinology and Diabetes Unit of University Campus Bio-Medico in Rome

ELIGIBILITY:
Inclusion Criteria:

* T1D patients
* aged 17-50 years
* disease duration > 1 year
* BMI >25

Exclusion Criteria:

* learning disabilities
* presence of chronic conditions potentially able to influence daily activities (visual or auditory disability, motor impairment for neurological or orthopaedic problems).
* T1D patients affected from diabetic complications
* pregnancy

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
efficacy of DCI oral supplementation on metabolic control | 6 months
  efficacy of DCI oral supplementation on metabolic control as assessed by HbA1c (%)

SECONDARY OUTCOMES:
BMI kg/m2 | 6 months
  reduction of BMI
Insulin Requirement (I.R.) IU/kg | 6 months
  reduction of I.R.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pozzilli, MD, Principal Investigator — University Campus Bio-medico
Locations (1):
- University Campus Bio Medico, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maurizi AR, Menduni M, Del Toro R, Kyanvash S, Maggi D, Guglielmi C, Pantano AL, Defeudis G, Fioriti E, Manfrini S, Pozzilli P. A pilot study of D-chiro-inositol plus folic acid in overweight patients with type 1 diabetes. Acta Diabetol. 2017 Apr;54(4):361-365. doi: 10.1007/s00592-016-0954-x. Epub 2016 Dec 30. PMID 28039583